CLINICAL TRIAL: NCT03136419
Title: Microbiota and Immune microEnvironment in Pouchitis: Randomized Controlled Trial Oral Administration of Lactobacillus Casei DG After Ileostomy Closure in Ileal Pouch Mucosa
Brief Title: Microbiota and Immune microEnvironment in Pouchitis
Acronym: MEP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Imerio Angriman, Assistant Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEP1
Record Dates: First submitted 2017-04-05; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pouchitis; Ulcerative Colitis; Ileal Pouch
Keywords: microbiota; innate immunity
MeSH Terms: conditions — Pouchitis; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo capsules bis in die for 8 weeks
  Interventions: Dietary Supplement: Placebo
- Experimental (Experimental): Lactobacillus casei DG capsules bis in die for 8 weeks
  Interventions: Dietary Supplement: Lactobacillus casei DG

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei DG — Lactobacillus casei DG probiotic supplementation for 8 weeks
  Arms: Experimental
Dietary Supplement: Placebo — Placebo supplementation for 8 weeks
  Arms: Control

SUMMARY:
Microbiota and innate immunity in pouchitis: predisposing factors and modulation of the inflammation with probiotics.

Around 20-25% of ulcerative colitis patients undergo restorative proctocolectomy with ileal pouch anal anastomosis. Pouchitis is an idiopathic inflammatory disease that may occur in ileal pouches. In our recent studies, we showed altered microbiota and innate immunity relationships in pouchitis. We plain to perform a double-blind, placebo-controlled trial probiotic therapy vs placebo starting at the time of ileostomy closure to evaluate the impact of microbiota that colonizes the pouch mucosa in the pathogenesis of pouchits, to determine how expression and activation status of the innate immunity system in different cell types and anatomical districts of pouch mucosa relate to microbiota population and follow-up the clinical outcome of anal pouches in light of microbiota-innate immune system interplay.

Our study will include three phases:

1. analysis of the intestinal microbiota with High Throughput Sequencing Unit and anaerobes cultures
2. characterization of innate immunity with TLR, NLR, nicotinic receptors and LPMC analysis
3. assessment of microbiota and innate immune system in the ileal pouch before ileostomy closure, 2 months after ileostomy closure and after 1 year follow up.

DETAILED DESCRIPTION:
Study aims

The working hypothesis is that a disruption of gut microbiota homeostasis, either spontaneous or caused by the deregulation of the innate immunity machinery within the pouch mucosa, contributes to the onset of chronic/relapsing pouchitis. Taking into account that bacterial colonization of the pouch mucosa can be ideally studied since its generation, this can be considered as an ideal model to study the interplay between gut microbiota and innate immune system. Therefore, the goal of this Research Unit is to establish how dysbiosis and innate immunity machinery dysfunction are established and how this disfunction contributes to the onset and maintenance of pouchitis. To address these relevant pathophysiological issues in light of their therapeutic implications, we plan to perform a randomized double-blind study probiotics vs placebo in patients who will undergo colectomy and subsequent ileal pouch-anal anastomosis to enrolling the patients at the time of ileostomy colure to:

1. evaluate composition and pathogenic properties of the microbiota that colonizes the pouch mucosa after ileostomy closure;
2. determine how expression and activation status of the innate immunity system in different cell types and anatomical districts of pouch mucosa relate to ileostomy closure;
3. follow-up the clinical outcome of anal pouches in light of microbiota-innate immune system interplay.

Study design In a two year period we calculated to enrol at least 32 patients who will be randomized at ileostomy closure in a group receiving placebo (16 patients) and in a group receiving lactobacillus casei GD oral supplementation for 8 weeks (16 patients). Mucosa samples will be harvested at ileostomy closure and at pouch endoscopy at 8 weeks and at 12 months.We will consider eligible candidates all patients with UC who will undergo restorative proctocolectomy with ileal pouch anal anastomosis and that will attend our outpatient's clinic for routine endoscopic and clinical follow-up. Patients with cuffitis (inflammation of the rectal mucosa remnant) or Crohn's disease of the pouch (with perianal fistulae or with inflammation of the afferent ileal limb), as well as patients who will have received antibiotic or probiotic therapy during the previous 30 days will be excluded from the study. Patients with PDAI>7 will be considered as overt pouchitis. The protocol will comply with the principles of the amended Declaration of Helsinki.

Each patient will be provided with detailed information about the study aims and methodology and will be asked to give written, informed consent prior to enrolment. During this period patients will be asked to undergo pouch endoscopy with mucosal biopsies, faecal and blood sampling at three following time: a) before ileostomy closure, b) 2 months after ileostomy closure, c) 12 months after ileostomy closure (or before, in case of overt pouchitis). Based on clinical, endoscopic and histological criteria and PDAI we will assess the disease severity [5]. Based on histological and endoscopic acute inflammation as well as clinical symptoms, patients with a total PDAI >7 will be classified as having acute pouchitis.

Endoscopy of the pouch will be performed without sedation. The afferent loop, the pouch will be carefully examined and biopsy sampling will be performed: two samples for microbiota characterization, two for conventional histology, four for molecular biology and cytofluorimetric analysis. Biopsies will be handled and stored accordingly to the different studies.

Microbiota assessment:

To characterize bacteria adherent to the pouch mucosa biopsies from the ileal pouch will be either immediately gently washed to remove loosely adherent microbes and then frozen in liquid nitrogen for subsequent DNA extraction, or placed in thioglycolate medium to preserve anaerobic microbes for subsequent cultures.

Relative abundance of bacterial phyla in faecal specimens will be estimated by sequencing the PCR amplicons targeting 16S rRNA gene for the DNA samples extracted from each faecal specimen. PCR will be performed using the primer set (784F: 5′-AGGATTAGATACCCTGGTA-3′ and 1061R: 5′-CRRCACGAGCTGACGAC-3′) that targets the V5-V6 region of the 16S rRNA genes [38]. To amplify the targeted region, 1 μl of extracted DNA will serve as template in 50-μl reactions using Prime STAR HS premix (Takara Bio Inc., Japan). Products of the two reconditioning PCR reactions per sample will be combined and purified using QIAquick PCR purification columns (Qiagen). The amplified PCR products will be used as a template for pyrosequencing with the GS Junior platform (454 Life Sciences). Pyrosequencing will be performed by following the manufacturer's instruction using MID tags. We expect to obtain about 15,000 sequencies for each sample, on the average. The obtained data will be subjected to a data analysis performed by computational tools. Bacterial rRNA typing will be performed by BLASTN search against the comprehensive rRNA database "silva" release 94 [39] using a threshold of E-value <1E-40. All the bacterial species obtained from each faecal sample will be classified into their phylogenetic groups and the proportion of different phyla will be estimated. The estimation of operational taxonomic unit (OTU) will be performed by the program ESPRIT using default settings [40].

For microbiological cultures biopsies immediately placed in thioglycolate medium (to protect anaerobic microbes from oxygen exposure) will be further manipulated in an anaerobic hood filled with C02:H2 (95:5) atmosphere. Biopsies will be washed in sterile dye-gassed saline solution supplemented with 0.016% dithioerythritol to remove the mucus and following cell hypotonic lysis in sterile water, seeded in proper agar plates to evaluate the superficial microflora. [35]. Samples will be seeded on non-selective (Brain Heart Infusion Agar, BHA) and selective media for Enterobacteriacae spp (MacConkey agar) and Lactobacillus spp (Rogosa SL agar).

BHA and MacConkey agar plates will be cultured in anaerobic and aerobic conditions (24 and 72 hrs, respectively), while Rogosa SL Agar plates will be only cultured in anaerobic conditions (72 hrs) at 37°C. Colonies will be counted, grouped on the basis of morphological appearance and subjected to morphological analysis by Gram staining (Biolife S.r.l.). Then microbes will be subjected to molecular characterization, performed by sequencing of PCR amplicons of 16S rRNA using an "Abi Prism TM Big Dye TM Terminator Cycle Sequencing Ready Reaction Kit" [24]. Isolates will be further characterized according to their pathogenicity potential (i.e. toxigenic profile and antibiotic resistance).

Mucosal innate immune environment

Analysis of the inflammatory network in the pouch mucosa will include

1. quantification of cytokines [IL-1ß, IL-6, TNF- , TGF ß, IL-10 and IL-4 and chemokines [MCP1,] level by Bio-Plex cytokine immunoassay. One biopsy will be homogenated and the clear supernatant used for the contemporary quantification of multiple cytokines and chemokines by custom-designed assays;
2. analysis of TLRs network (mRNA quantification and protein distribution) by quantitative RT-PCR and immunohistochemistry, respectively;
3. assessment of activation status of macrophages, dendritic cells, infiltrating lymphocytes evaluating surface markers (i.e.) and intracellular cytokines pattern (i.e. TNF , IFN , IL4, IL10) by cytofluorimetric analysis. Two biopsies will be subjected to gentle enzymatic digestion and then stained with properly labelled antibodies directed against surface antigens or intracellular cytokines.

Mucosal anti-microbial activity. To characterize the anti-bacterial peptide-network in the pouch mucosa responsible to shape-up the adherent microbiota we will a) determine the anti-microbial properties of mucosal extracts by performing in vitro anti-bacterial toxicity assay [37]; b) quantify epithelial and leucocytes-derived anti-microbial defensins (such as Def2, Def3; DEFA5; DEFA6) by quantitative RT-PCR.

Histological evaluation:

For routine histological examination two biopsies will be fixed in 4% PFA for 24 Hrs, then dehydrated and embedded in paraffin, and sections (5 μm thick) will be cut and subjected to standard haematoxylin/eosin (H&E) stain. To quantify inflammatory severity will be used the Floren et al. score [41].

Systemic and intestinal inflammation assessment

Systemic and local inflammatory state will be assessed at each experimental timeline by: erythrocyte sedimentation rate (ESR), white blood cell count (WBC), platelets blood count (PLT), CRP and fecal lactoferrin, respectively. ESR will be measured by the Westergren method. CRP will be detected by immuno-nephelometry (normal: <6 mg/l; pathological >6mg/l). Total protein and albumin will be assessed with the biuret method. WBC, platelets counts and haemoglobinaemia will be obtained with standard full blood cell count. Fecal lactoferrin will be dosed by an ELISA test that uses rabbit polyclonal antibodies specific for human lactoferrin on frozen stool samples.

Statistical analysis

Statistical analysis will be performed using Windows Microsoft Excel and a Statistica 7.1 (Statsoft, Inc.) software. Continuous data will be expressed as median (range); dichotomic data will be expressed as frequency and proportion. Non-parametric tests will be used. Correlation between bacteria strains and inflammatory parameters will be calculated with Spearman test to evaluate the etio-pathogenetic role of each strain. Relevant correlation coefficient will be not inferior to 0.50 and, setting a two-tails statistic significance level at 0.05 and power at 0.20, the consequent sample size will have to be at least of 29 patients. Comparison between pouchitis and healthy pouch will be performed with Mann-Whitney U test. Set a level of statistical significance at 0.05 and a power at 0.20 the consequent sample size required for comparison will be 16 patients for each group. In conclusion at least 32 patients will be enrolled in this study. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

All patients with UC who will undergo restorative proctocolectomy with ileal pouch anal anastomosis and that will attend our outpatient's clinic for routine endoscopic and clinical follow-up.

Exclusion Criteria:

Patients with cuffitis (inflammation of the rectal mucosa remnant) or Crohn's disease of the pouch (with perianal fistulae or with inflammation of the afferent ileal limb), as well as patients who will have received antibiotic or probiotic therapy during the previous 30 days will be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
quantification of inflammatory cytokines in the ileal mucosa levels by Bio-Plex cytokine immunoassay | 8 weeks
  IL-1ß, IL-6, TNF-alpha

SECONDARY OUTCOMES:
quantify epithelial and leucocytes-derived anti-microbial defensins | 8 weeks
  Def2, Def3; DEFA5; DEFA6 by quantitative RT-PCR
pouchitis episodes | 12 months
  pouchitis episodes evaluated at PDAI >5
Relative abundance of bacterial phyla in faecal specimens | 8 weeks
  Relative abundance of bacterial phyla in faecal specimens will be estimated by sequencing the PCR amplicons targeting 16S rRNA gene for the DNA samples extracted from each faecal specimen.
Systemic and local inflammatory status | 12 months
  Systemic and local inflammatory state will be assessed at each experimental timeline by: erythrocyte sedimentation rate (ESR), white blood cell count (WBC), platelets blood count (PLT), CRP and fecal lactoferrin
Histological inflammatory severity | 8 weeks
  Floren score
activation status of macrophages, dendritic cells, infiltrating lymphocytes | 8 weeks
  assessment of activation status of macrophages, dendritic cells, infiltratinglymphocytes evaluating surface markers (i.e.) and intracellular cytokines pattern (i.e. TNF , IFN , IL4, IL10) by cytofluorimetric analysis.
analysis of TLRs network | 8 weeks
  quantitative RT-PCR and immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Imerio Angriman, MD, Principal Investigator — University of Padova
Locations (1):
- Imerio Angriman, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Angriman I, Scarpa M, Castagliuolo I. Relationship between pouch microbiota and pouchitis following restorative proctocolectomy for ulcerative colitis. World J Gastroenterol. 2014 Aug 7;20(29):9665-74. doi: 10.3748/wjg.v20.i29.9665. PMID 25110406
- [Result] Scarpa M, Grillo A, Scarpa M, Brun P, Castoro C, Pozza A, Cavallo D, Faggian D, Ruffolo C, D'Inca R, Bardini R, Castagliuolo I, Angriman I. Innate immune environment in ileal pouch mucosa: alpha5 defensin up-regulation as predictor of chronic/relapsing pouchitis. J Gastrointest Surg. 2012 Jan;16(1):188-201; discussion 201-2. doi: 10.1007/s11605-011-1720-6. Epub 2011 Oct 8. PMID 21983950
- [Result] Scarpa M, Grillo A, Pozza A, Faggian D, Ruffolo C, Scarpa M, D'Inca R, Plebani M, Sturniolo GC, Castagliuolo I, Angriman I. TLR2 and TLR4 up-regulation and colonization of the ileal mucosa by Clostridiaceae spp. in chronic/relapsing pouchitis. J Surg Res. 2011 Aug;169(2):e145-54. doi: 10.1016/j.jss.2011.04.003. Epub 2011 May 5. PMID 21601883
- [Result] Scarpa M, Grillo A, Faggian D, Ruffolo C, Bonello E, D'Inca R, Scarpa M, Castagliuolo I, Angriman I. Relationship between mucosa-associated microbiota and inflammatory parameters in the ileal pouch after restorative proctocolectomy for ulcerative colitis. Surgery. 2011 Jul;150(1):56-67. doi: 10.1016/j.surg.2011.02.009. Epub 2011 May 5. PMID 21549404
- [Result] Scarpa M, Mescoli C, Rugge M, D'Inca R, Ruffolo C, Polese L, D'Amico DF, Sturniolo GC, Angriman I. Restorative proctocolectomy for inflammatory bowel disease: the Padova prognostic score for colitis in predicting long-term outcome and quality of life. Int J Colorectal Dis. 2009 Sep;24(9):1049-57. doi: 10.1007/s00384-009-0700-8. Epub 2009 Apr 22. PMID 19415309
- [Derived] Angriman I, Scarpa M, Savarino E, Patuzzi I, Rigo A, Kotsafti A, Stepanyan A, Sciuto E, Celotto F, Negro S, Caruso A, Ruffolo C, Bardini R, Pucciarelli S, Barberio B, Spolverato G, Zingone F, D'Inca R, Castagliuolo I, Scarpa M. Oral administration of Lactobacillus casei DG(R) after ileostomy closure in restorative proctocolectomy: a randomized placebo-controlled trial (microbiota and immune microenvironment in pouchitis -MEP1). Gut Microbes. 2024 Jan-Dec;16(1):2423037. doi: 10.1080/19490976.2024.2423037. Epub 2024 Nov 1. PMID 39485259